CLINICAL TRIAL: NCT06509880
Title: The Role of Neutrophil Mitochondrial Dysfunction in Medical Rehabilitation During Palliative Chemotherapy for Metastatic Colorectal Cancer
Brief Title: Immunosurveillance for Metastatic Colorectal Cancer
Acronym: ISMCC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MIPO Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2024-07-06; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Monitoring, Immunologic
Keywords: Colorectal Cancer; Chemotherapy; Rehabilitation; Mitochondria; Sodium Nucleinate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sodium nucleinate; Folfox protocol

STUDY DESIGN:
Intervention Model Description: The goal of this study type: clinical trial is to primary purpose: e.g., learn if intervention or health behavior can treat, prevent, diagnose etc. and improve the quality of life and reduce one-year mortality in palliative treatment of metastatic forms of colorectal cancer.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients were randomized into two groups - main and control - using the envelope method. No surnames were indicated on the medical records. The researcher did not know to which group the patient would fall. The nurse did not know which group the patient was in when carrying out medical appointments. The physician-researcher was from another clinic and even from another city, who performed the laboratory analysis did not know the age, sex or diagnosis of the patient who was identified from the envelope. The social worker was from another clinic and when processing the results of the quality of life tests did not know to whom they belonged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy according to the FOLFOX regimen in combination with sodium nucleonate (Active Comparator): Рatients with metastatic colorectal cancer (stages T3-4 N1-2 M), receiving four courses of FOLFOX chemotherapy (Day 1-2: Oxaliplatin 100 mg/m2 IV infusion, given as a 120 minutes IV infusion in 500 mL D5W, concurrent with leucovorin 400 mg/m2 (or levoleucovorin 200 mg/m2) IV infusion, followed by 5-FU 400 mg/m2 IV bolus, followed by 46-hour 5-FU infusion (2400 mg/m2 for first two cycles, and may be increased to 3000 mg/m2 if tolerated by patient (no toxicity > grade 1 during the first two cycles), days 3-14: Rest days) combined with mitochondrial immunotherapy using sodium nucleinate. The medical rehabilitation protocol involved administering sodium nucleinate at 50 mg per day: 25 mg in the morning and 25 mg at lunch before meals, daily for four months.
  Interventions: Dietary Supplement: Adenorine; Drug: FOLFOX regimen
- Chemotherapy according to the FOLFOX regimen (Sham Comparator): Рatients with metastatic colorectal cancer (stages T3-4 N1-2 M), who received only four courses of FOLFOX chemotherapy (Day 1-2: Oxaliplatin 100 mg/m2 IV infusion, given as a 120 minutes IV infusion in 500 mL D5W, concurrent with leucovorin 400 mg/m2 (or levoleucovorin 200 mg/m2) IV infusion, followed by 5-FU 400 mg/m2 IV bolus, followed by 46-hour 5-FU infusion (2400 mg/m2 for first two cycles, and may be increased to 3000 mg/m2 if tolerated by patient (no toxicity > grade 1 during the first two cycles), days 3-14: Rest days). In both groups, general and biochemical blood analyses were conducted monthly
  Interventions: Biological: Placebo; Drug: FOLFOX regimen

INTERVENTIONS:
Dietary Supplement: Adenorine — The immunostimulating effect of the drug is associated with its ability to activate the cells of the monocyte-macrophage system, thus increasing the functional activity of all parts of the body, stimulating the repair and regeneration of cells and tissues. It reduces the symptoms of the iflammatory process, stimulates the development of granulations and growth of epithelial tissues, accelerates the process of cleansing and healing of infected wounds. While with healthy people, it can be used as a phylactic drug that improves immunity protection. It was proved that when the drug is used externally, activation of macrophages occurs, thus accelerating wound cleansing process and stimulating reparative processes. In cases when thermal injury to the skin is more than 15-20% of the surface, there is a "stress syndrome" that suppresses the immune system. When exposed to DNA-Na, lymphocyte activation occurs, wound cleansing processes are accelerated.
  Other Names: natural oligodeoxynucleotide; sodium nucleinate
  Arms: Chemotherapy according to the FOLFOX regimen in combination with sodium nucleonate
Biological: Placebo — Placebo
  Arms: Chemotherapy according to the FOLFOX regimen
Drug: FOLFOX regimen — (Day 1-2: Oxaliplatin 100 mg/m2 IV infusion, given as a 120 minutes IV infusion in 500 mL D5W, concurrent with leucovorin 400 mg/m2 (or levoleucovorin 200 mg/m2) IV infusion, followed by 5-FU 400 mg/m2 IV bolus, followed by 46-hour 5-FU infusion (2400 mg/m2 for first two cycles, and may be increased to 3000 mg/m2 if tolerated by patient (no toxicity > grade 1 during the first two cycles), days 3-14: Rest days)

SUMMARY:
The goal of this study type: clinical trial is to primary purpose: e.g., learn if intervention or health behavior can treat, prevent, diagnose etc. and improve the quality of life and reduce one-year mortality in palliative treatment of metastatic forms of colorectal cancer.. The main question[s] it aims to answer [is/are]:

1. Does the combination of sodium adenosine nucleonate and FOLFOX course affect chemotherapy efficacy and treatment adherence?
2. which of the assays can be considered a marker of the efficacy of the combination of sodium nucleonate and FOLFOX?
3. Effect of the combination of adenosine nucleonate sodium and FOLFOX on patient quality of life?

   * If there is a comparison group:_ Researchers will compare [compare the two arms of the main arm 100 patients and the control arm 100 patients] to see if [insert effects].

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

1. To evaluate the efficacy of palliative care with 4 courses of FOLFOX-based chemotherapy combined with sodium nucleonate for metastatic colorectal cancer (CRC) in the main group.
2. In the control group in metastatic colorectal cancer to study the efficacy of 4 courses of stand-alone standard chemotherapy according to the FOLFOX scheme.
3. To examine the obtained results and compare the quality of life, dynamics of laboratory tests and overall survival in the main and control groups.
4. To evaluate the influence of quantitative and qualitative indices of mitochondrial activity in the blood of patients in the main and control groups.
5. To reveal the correlation between the dynamics of mitochondrial dysfunction, quality of life of patients, tolerance to toxic effects of chemotherapy, as well as the reduction of one-year mortality in patients with colorectal cancer.

DETAILED DESCRIPTION:
Materials and methods of the study. According to the approved by the Local Ethical Committee of the Kazakh National Medical University, it was planned to include in the study 200 patients from 19 regions of Kazakhstan with histological, verified diagnosis of "colorectal cancer", treated in oncological centers of 4 regions of Kazakhstan, where there were University Clinics.

Distribution of Colorectal Cancer Patients (CRC) by Type of Treatment.

1. Main group - Chemotherapy according to the FOLFOX regimen in combination with sodium nucleonate 100
2. Control group Chemotherapy according to the FOLFOX regimen 100 Study Design The study design included an evaluation of the effectiveness of FOLFOX chemotherapy in combination with sodium nucleinate immunotherapy in 187 patients with metastatic colorectal cancer at stages T3-4 N1-2 M1. Randomization into two groups-main and control-was performed using the envelope method.

The main group included 89 patients with metastatic colorectal cancer (stages T3-4 N1-2 M), receiving four courses of FOLFOX chemotherapy combined with mitochondrial immunotherapy using sodium nucleinate. The medical rehabilitation protocol involved administering sodium nucleinate at 50 mg per day: 25 mg in the morning and 25 mg at lunch before meals, daily for four months.

The control group consisted of 98 patients with metastatic colorectal cancer (stages T3-4 N1-2 M), who received only four courses of FOLFOX chemotherapy. In both groups, general and biochemical blood analyses were conducted monthly.

Additionally, before the start of treatment and one month after the end of treatment, PET-CT scans were performed, levels of tumour markers CEA and CA-19-9 were determined, immunological status CD4/CD8 and mitochondrial activity of neutrophils were assessed, and echocardiography was conducted to determine the left ventricular ejection fraction. A well-being questionnaire (the European Organization for Research and Treatment of Cancer (EORTC) QLQ-CR29) was also administered.

Critical Points

1. Reduction in treatment interruptions due to leukopenia, neutropenia, and infectious complications during chemotherapy for metastatic colorectal cancer (CRC).
2. Increased percentage of tumour process stabilization during palliative chemotherapy for CRC.

Reduction in one-year mortality during palliative treatment of metastatic CRC. Statistical analysis of the study results was performed using the application program package "Statistica 7.0" for Windows (StatSoft, USA). The Mann-Whitney U-criterion was used to compare the studied samples by qualitative indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Oncological patients with a histologically confirmed diagnosis of "colorectal cancer" and regional metastases at stages T1-4 N1-2 M0, who have provided informed consent to participate in the study.
2. Oncological patients with a histologically confirmed diagnosis of "colorectal cancer" with distant metastases at stages T1-4 N1-2 M1, who have provided informed consent to participate in the study.

Exclusion Criteria:

1. Oncological patients with a histologically confirmed diagnosis of "colorectal cancer" and regional metastases at stages T1-4 N1-2 M1, who have active forms of pulmonary tuberculosis, decompensated diabetes, decompensated cardiac, vascular, lung, liver, and renal failure.
2. Oncological patients with a histologically confirmed diagnosis of "colorectal cancer" with regional and distant metastases at stages T1-4 N1-2 M1, who have not provided informed consent to participate in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-CR29 | before the start of treatment and one month after the end of treatment
  the European Organization for Research and Treatment of Cancer (EORTC) QLQ-CR29 max242 min59. whether higher scores mean a worse outcome
Dynamics of mitochondrial activity neutrophils | before the start of treatment and one month after the end of treatment
  Mitochondrial dynamics refers to the changing process of fission, fusion, mitophagy and transport, which is crucial for optimal function in signal transduction and metabolism. An imbalance in mitochondrial dynamics can disrupt mitochondrial function, leading to abnormal cellular fate, and a range of diseases, including neurodegenerative disorders, metabolic diseases, cardiovascular diseases and cancers. Herein, we review the mechanism of mitochondrial dynamics, and its impacts on cellular function. the normal range of cell distribution 30-60% 30% of the 200 cells counted. whether higher scores mean a better outcome.
Positron emission tomography/computed tomography | before the start of treatment and one month after the end of treatment
  Positron emission tomography (PET/CT) is used prior to surgery in patients with metastatic or recurrent colorectal cancer to identify those with potentially curable disease or to dynamically monitor the course of the disease. normally, it does not accumulate an isotope. whether higher scores mean a worse outcome.
CEA | before the start of treatment and one month after the end of treatment
  Carcinoembryonic Antigen Oncomarker is used in the diagnosis of malignant and benign tumors of GI organs or to dynamically monitor the course of the disease. normal concentration min=0 ng/ml max=5,5 ng/ml. whether higher scores mean a worse outcome.
CA 19-9 (Carbohydrate (carbohydrate) antigen 19-9) | before the start of treatment and one month after the end of treatment
  CA 19-9 was discovered in the early 1980s by researchers working to identify tumor antigens in colorectal cancer or to dynamically monitor the course of the disease. normal concentration min=0 U/ml, max=27,0 U/ml. whether higher scores mean a worse outcome.
CD4/ CD8 ratio | before the start of treatment and one month after the end of treatment
  Prognostic value of the CD4+/CD8+ ratio of tumour infiltrating lymphocytes in colorectal cancer. The normal range of CD4+/CD8+ is from 1.0 to 4.0. the ratio level above and below the norm is considered a bad prognostic sign

SECONDARY OUTCOMES:
Echocardiography with determination of left ventricular ejection fraction | before the start of treatment
  Echocardiography with determination of left ventricular ejection fraction to detect impaired function of vital organs as a factor of exclusion from the study group. in the case of a violation of the vital function of the heart below normal parameters, it is a negative sign and the patient is subject to exclusion from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- MIPOClinic, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No